CLINICAL TRIAL: NCT03757611
Title: A 12 Week, Multi-center, Randomized, Double-blind, Placebo-controlled Clinical Trial for the Evaluation of the Efficacy and Safety of Tabetri on Osteoarthritis
Brief Title: Efficacy and Safety of Tabetri on Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Collaborators: Nutribiotech Co., Ltd. (Industry); Neonutra (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: JS-CT-2017-02
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tabetri (Experimental): Tabetri capsule will be administered orally twice daily for 12 weeks
  Interventions: Dietary Supplement: Tabetri capsule
- Placebo (Placebo Comparator): Placebo capsule will be administered orally twice daily for 12 weeks
  Interventions: Dietary Supplement: Placebo capsule

INTERVENTIONS:
Dietary Supplement: Tabetri capsule — 1,000 mg/capsule (Taheebo extract 600 mg/day)
  Arms: tabetri
Dietary Supplement: Placebo capsule — 1,000 mg/capsule
  Arms: Placebo

SUMMARY:
This study is a 12-week, multicenter, randomized, double-blind, placebo-controlled clinical trial in order to evaluate the efficacy and safety of tabetri on osteoarthritis.

DETAILED DESCRIPTION:
This study is prospectively conducted to investigate the efficacy and safety of tabetri in patients diagnosed with osteoarthritis at 4 locations of Jaseng Hospital of Korean Medicine (Gangnam, Haeundae, Daejeon, and Bucheon).

ELIGIBILITY:
Inclusion Criteria:

* Male or female 40 ~ 75 years of age
* VAS (Visual Analogue Scale) over 30mm
* Kellgren & Lawrence Grade I~II by X-ray
* Subject who agrees to participate in this clinical trial by themselves and signs the Informed Consent Form (ICF)

Exclusion Criteria:

* Subjects who diagnosed inflammatory arthritis (rheumatoid arthritis, fibromyalgia, systemic lupus erythematosus, septic arthritis, gout)
* Joint space under 2 mm by X-ray
* Kellgren & Lawrence Grade over III with osteophyte, irregularly-shaped auricular surfaces, or subchondral bone cyst by X-ray
* Subjects who diagnosed cardiovascular disease, immune disease, infectious diseases, tumor diseases
* Subjects having gastrointestinal diseases
* Uncontrolled hypertension patients (Blood pressure ≥ 160/100mmHg)
* Uncontrolled diabetes mellitus patients (fasting glucose level ≥ 180mg/dl)
* Patients with TSH <= 0.1 uIU/mL or >= 10 uIU/mL
* Subjects have attended abnormal values at AST or ALT (3 times excess at upper limit of the normal values)
* Subjects have attended abnormal values at creatinine (2 times excess at upper limit of the normal values)
* Pregnancy, breast-feeding, or subjects who have a plan to pregnancy within 3 months
* Use of osteoarthritis treatment drugs or dietary supplements within 2 weeks prior to screening
* Psychiatric disorder patient (schizophrenia, depressive disorder, drug abuse)
* History of osteoarthritis treatment therapy within 2 weeks prior to screening
* Have participated in another clinical trial within the 3 months prior to screening
* Subjects who have hypersensitivity history about investigational product
* Have difficulty to be participated in this clinical trial by investigator's decision

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
VAS (Visual Analogue Scale) | Change of the week 6 and 12 from baseline
  VAS is used to measure changes in joint pain on 6 and 12 weeks after administration in comparison with baseline. It is presented as a 100-mm horizontal line on which the patient's pain intensity is presented by a point between the extremes of "no pain at all" and "worst pain imaginable."
K-WOMAC (Korean-Western Ontario and McMaster Universities) | Change of the week 6 and 12 from baseline
  K-WOMAC is used to measure changes in joint pain and function on 0, 6, and 12 weeks after administration in comparison with baseline. It measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68).
KSF-36 (Korean-Short Form Health Survey 36) | Change of the week 6 and 12 from baseline
  KSF-36 is used to measure changes in physical and mental function on 0, 6, and 12 weeks after administration in comparison with baseline. It is a 36-item self-report measure designed to assess health-related functioning. It contains eight subscales with four pertaining to physical functioning and four pertaining to psychological functioning. Scores on each subscale can range from 0 to 100, with a higher score representing better health-related functioning. Two composite scores are calculated by averaging all of the scores for four subscales pertaining to each of the two general aspects of functioning.

SECONDARY OUTCOMES:
Subject's global impression of change scale | 6 and 12 weeks
  The change in activity limitations, symptoms, emotions and overall quality of life, related to painful condition that is assessed by subject
  Level of Quality
  * Excellent (category 1): substantial overall improvement of symptoms
  * Good (category 2): overall improvement of symptoms
  * Neutral (category 3): no change compared with before
  * Worse (category 4): overall deterioration of symptoms
  * Very much worse (category 5): substantial overall deterioration of symptoms
Investigator's global impression of change scale | 6 and 12 weeks
  The change in activity limitations, symptoms, emotions and overall quality of life, related to painful condition that is assessed by investigator
  Level of Quality
  * Excellent (category 1): substantial overall improvement of symptoms
  * Good (category 2): overall improvement of symptoms
  * Neutral (category 3): no change compared with before
  * Worse (category 4): overall deterioration of symptoms
  * Very much worse (category 5): substantial overall deterioration of symptoms
ESR (Erythrocyte sedimentation rate) | Change of the week 12 from baseline
  ESR to measure changes in blood inflammatory marker on 12 weeks after administration in comparison with baseline
CRP (C-reactive protein) | Change of the week 12 from baseline
  CRP to measure changes in blood inflammatory marker on 12 weeks after administration in comparison with baseline

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, KMD, MPH, Principal Investigator — Jaseng Medical Foundation
Locations (4):
- South Korea (4):
  - Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si, Gyeonggi-do
  - Haeundae Jaseng Hospital of Korean Medicine, Busan
  - Daejeon Jaseng Hospital of Korean Medicine, Daejeon
  - Jaseng Hospital of Korean Medicine, Seoul

IPD SHARING:
Plan to Share IPD: Undecided